CLINICAL TRIAL: NCT04493827
Title: Distribution and Prognostic Impact of Oncogenic Drivers in Metastatic Lung Adenocarcinoma : a Retrospective Monocentric Study in Nancy University Hospital Center
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2019PI224
Record Dates: First submitted 2020-06-29; First posted 2020-07-30 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-06

CONDITIONS: Adenocarcinoma of Lung Stage IV; Adenocarcinoma of Lung, Response to Tyrosine Kinase Inhibitor in, Somatic
MeSH Terms: conditions — Adenocarcinoma of Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The recent discovery of oncogenic drivers has revolutionized the management of advanced lung cancer by development of tyrosine kinase inhibitors targeted therapies. Prevalence of daily tobacco use is evaluated at 31,3 % in Grand-Est region, the only French region with a statistically significative difference for smoking habits. This region shows a higher incidence (+ 13 %) and mortality for lung cancer in comparison to the average for other French regions. The objectives of our studie were to estimate the distribution of oncogenic drivers and analyse their prognostic impacts in the Nancy University Hospital Center metastatic lung adenocarcinoma's population.

ELIGIBILITY:
Inclusion Criteria:

* Lung adenocarcinoma
* Patients diagnosed at a metastatic stage
* Patient who benefited an oncogenic driver research on their histologic samples
* Medical follow-up entirely done in Nancy Central Hospital

Exclusion Criteria:

* Patients with double histology
* Synchronous cancer
* Patients with surgical care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic lung adenocarcinoma diagnosed between 2012 and 2014 with a medical follow-up entirely done in Nancy Central Hospital
Sampling Method: Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Overall survival | over a period of 5 years (Day 0 = anatomopathological diagnosis)
  Time (in months) from anatomopathological diagnosis to death
Progression Free survival | over a period of 5 years (Day 0 = anatomopathological diagnosis)
  Time (in months) from anatomopathological diagnosis to progression of the disease assessed by RECIST criteria
Distribution in percentage of main oncogenic drivers in histological samples from metastatic lung adenocarcinoma | At base line (Day 0 = anatomopathological diagnosis)
  Distribution in percentage of main oncogenic drivers (KRAS, EGFR, ALK, ROS-1, BRAS and HER2), assessed by Sanger sequencing or FISH method in histological samples from metastatic lung adenocarcinomas

SECONDARY OUTCOMES:
Distribution in percentage of metastasis sites according oncogenic drivers | At baseline (Day 0 = anatomopathological diagnosis)
  Distribution in percentage of metastatic sites assessed by CT-scan for metastatic lung adenocarcinomas according oncogenic drivers (KRAS, EGFR, ALK, ROS-1, BRAS and HER2)

CONTACTS AND LOCATIONS:
Overall Officials: Angelica Tiotiu, Study Director — Nancy Central Hospital
Locations (1):
- Centre Hospitalier Régional Universitaire, Vandœuvre-lès-Nancy, Meurthe Et Moselle, France